CLINICAL TRIAL: NCT04162834
Title: Effect of Papaverine on Intraoperative Renal Artery Blood Flow Volume in Patients Undergoing Robot-assisted Partial Nephrectomy : a Randomized, Placebo-controlled Study
Brief Title: Effect of Papaverine on Renal Artery Blood Flow Volume
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, MD, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20191111
Record Dates: First submitted 2019-11-10; First posted 2019-11-14 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Papaverine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papaverine group (Experimental): Immediately after the renal artery declamping, papaverine 30 mg (1 ample, 1 ml) is mixed with 5 ml of normal saline (total 6 ml) and sprinkled around the renal artery.
  Interventions: Drug: Papaverine
- Normal saline group (Active Comparator): Immediately after the renal artery declamping, normal saline 6 ml is sprinkled around the renal artery.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Papaverine — Immediately after the renal artery declamping, papaverine 30 mg (1 ample, 1 ml) is mixed with 5 ml of normal saline (total 6 ml) and sprinkled around the renal artery.
  Arms: Papaverine group
Drug: Normal saline — Immediately after the renal artery declamping, normal saline 6 ml is sprinkled around the renal artery.
  Arms: Normal saline group

SUMMARY:
The purpose of this study is to evaluate the effect of papaverine on renal artery blood flow after declamping of renal artery.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of papaverine on renal artery blood flow after declamping of renal artery in patients undergoing robot assisted partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with kidney cancer.
* Patients undergoing robot assisted partial nephrectomy under general anesthesia
* 20 years old ≤ age <80 years old
* Patients who voluntarily agreed to this clinical study
* eGFR ≥ 60 ml / min / 1.73 m2 (Chronic Kidney Disease Epidemiology Patients with Collaboration)

Exclusion Criteria:

* The tumor ≥ 7 cm in size
* Multiple renal mass
* If the surgery plan is changed due to open
* When surgery is performed together with other surgery
* Multiple renal artery
* Patients with hypersensitivity to papaverine
* Patients with atrioventricular block
* Pregnant and lactating women
* Patients using levodopa
* Refusal of patient

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Renal artery blood flow | at 2 minutes after papaverine administration
  Renal artery blood flow 2 minutes after papaverine administration by doppler sonography

SECONDARY OUTCOMES:
estimated glomerular filtration rate | at postoperative day 0
  estimated glomerular filtration rate using KIDGO equation
estimated glomerular filtration rate | at postoperative day 1
  estimated glomerular filtration rate using KIDGO equation
estimated glomerular filtration rate | at postoperative day 4
  estimated glomerular filtration rate using KIDGO equation
estimated glomerular filtration rate | at postoperative day 14
  estimated glomerular filtration rate using KIDGO equation
estimated glomerular filtration rate | at postoperative month 3
  estimated glomerular filtration rate using KIDGO equation
glomerular filtration rate using renal scan | at postoperative month 3
  glomerular filtration rate using renal scan

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD,PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No